CLINICAL TRIAL: NCT02419560
Title: Multi-institution Phase I/Ib Study of Ibrutinib With ABT-199 in Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Optimal Dose Finding Study ABT-199 and Ibrutinib in MCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig Portell, MD (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Craig Portell, MD, Assistant Professor of Medicine, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17983; ABT199-MCL-UVA-001 (Other: University of Virginia)
Record Dates: First submitted 2015-03-06; First posted 2015-04-17 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma, Mantle-Cell; Recurrent Lymphoma, Mantle-Cell
Keywords: Relapsed; Laboratory biomarker research; Pharmacologic study; Bruton's tyrosine kinase inhibitor; BCL-2 inhibitor
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — venetoclax; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT-199 and Ibrutinib Combination (Experimental): Participants will take ABT-199 (dose 100-400 mg) and Ibrutinib (dose 280-560 mg).
  Interventions: Drug: ABT-199 and Ibrutinib Combination

INTERVENTIONS:
Drug: ABT-199 and Ibrutinib Combination — Both are administered orally once daily.
  Other Names: GDC-0199; venetoclax; PCI-32765

SUMMARY:
The purpose of this study is to determine the optimal dosing scheme for the combination of ibrutinib with ABT-199 for the treatment of relapsed or refractory mantle cell lymphoma (MCL).

DETAILED DESCRIPTION:
This is a multi-center, study which will be open at up to 4 clinical sites. The purpose of this study is to determine the optimal dosing scheme for the combination of ibrutinib with ABT-199 for the treatment of relapsed or refractory mantle cell lymphoma (MCL). The main criterion for eligibility is MCL with measurable disease which is relapsed or refractory to at least 1 chemotherapy-containing regimen and has not been previously treated with ibrutinib.

This dose finding study will use a continual reassessment method, which accounts for both toxicity and efficacy in combinations of agents, to determine the optimal combination of the approved treatment ibrutinib with the investigational agent ABT-199. This study will accrue patients in two stages. In the initial stage, subjects will be accrued to dosing cohorts of increasing dosages of ABT-199 in combination with ibrutinib. The modeling is initiated once 1 subject experiences a dose limiting toxicity (DLT). During the modeling stage, treatment assignments will be made based on model prediction.

Subjects will remain on treatment until progression or unacceptable toxicity, and will be monitored for safety during the treatment interval. Safety will be evaluated by incidence of adverse events and number of discontinuations due to AEs. Efficacy endpoints include Overall Response Rate (ORR), Complete Response Rate (CRR), minimal residual disease response rate, and survival (PFS and OS). The study will also include exploratory analysis of the gene expression pattern in subjects who progress on treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Mantle Cell Lymphoma and has had at least one chemotherapy.
2. Subjects must have measurable or evaluable disease.
3. ECOG Performance Status of 0-2.
4. Must be referred for treatment with ibrutinib.
5. Must have adequate organ function.

Exclusion Criteria:

1. Subject is pregnant.
2. Prior malignancy (except nonmelanomatous skin cancer) unless disease free for a minimum of 2 years; non-invasive conditions such as carcinoma in situ of the breast, oral cavity, or cervix are all permissible.
3. Known CNS lymphoma.
4. Prior or current treatment with certain medications. Talk to Study Contact for specifics.
5. Subject is at high risk for TLS.
6. Subject has malabsorption syndrome or other condition which may affect an enteral route of administration.
7. Subject has known contraindication or allergy to both xanthine oxidase inhibitors and rasburicase.
8. Significant history of heart disease.
9. Subject has an active infection.
10. Known active Hepatitis B or Hepatitis C.
11. A serious uncontrolled medical disorder that in the opinion of the investigator would impair the ability of the subject to receive protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | 30 Days Following Start of Treatment

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events | Through 30 Days Following the Last Treatment
Overall Response Rate | Every Year Until Death; an Average of 2 Years
Complete Response Rate | Every Year Until Death; an Average of 2 Years
Progression-Free Survival | Every Year Until Death; an Average of 2 Years
Overall Survival | Every Year Until Death; an Average of 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Portell, MD, Study Chair — University of Virginia
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Jayappa KD, Tran B, Gordon VL, Morris C, Saha S, Farrington CC, O'Connor CM, Zawacki KP, Isaac KM, Kester M, Bender TP, Williams ME, Portell CA, Weber MJ, Narla G. PP2A modulation overcomes multidrug resistance in chronic lymphocytic leukemia via mPTP-dependent apoptosis. J Clin Invest. 2023 Jul 3;133(13):e155938. doi: 10.1172/JCI155938. PMID 37166997
- [Derived] Portell CA, Wages NA, Kahl BS, Budde LE, Chen RW, Cohen JB, Varhegyi NE, Petroni GR, Williams ME. Dose-finding study of ibrutinib and venetoclax in relapsed or refractory mantle cell lymphoma. Blood Adv. 2022 Mar 8;6(5):1490-1498. doi: 10.1182/bloodadvances.2021005357. PMID 34700344